CLINICAL TRIAL: NCT00470379
Title: Transcutaneous (Topical) Peptide Immunization With NY-ESO-1b (SLLMWITQC) Peptide Using Resiquimod as an Immune Adjuvant: A Pilot Study
Brief Title: Vaccine Therapy and Resiquimod in Treating Patients With Stage II, Stage III, or Stage IV Melanoma That Has Been Completely Removed by Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0578; P30CA015083 (NIH); MC0578 (Other: Mayo Clinic Cancer Center); 169-06 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — resiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunization with NY-ESO-1b (Experimental): Efficacy of maximal dose of topical resiquimod as immune adjuvant to intradermally administered NY-ESO-1b peptide vaccine.
  Interventions: Drug: resiquimod

INTERVENTIONS:
Drug: resiquimod — Escalating the dose of resiquimod applied to a fixed area of skin followed by application of topical NY-ESO-1b.

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Giving vaccine therapy together with resiquimod may make a stronger immune response and prevent or delay the recurrence of cancer.

PURPOSE: This clinical trial is studying the side effects, best dose, and best way to give vaccine therapy together with resiquimod in treating patients with stage II, stage III, or stage IV melanoma that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and immunization efficacy of the NY-ESO-1b peptide vaccine with resiquimod adjuvant in patients with completely resected stage II-IV melanoma.
* Collect, preliminarily, descriptive data on the impact of this regimen on time to melanoma relapse in these patients.

OUTLINE: This is a 3-step pilot, dose-escalation study of resiquimod.

* Step 1: Patients receive NY-ESO-1b peptide vaccine intradermally and topical resiquimod on day 1.

A cohort of 3-6 patients receives a maximal dose of resiquimod with NY-ESO-1b peptide vaccine.

* Step 2: Patients receive topical NY-ESO-1b peptide vaccine and topical resiquimod on day 1.

Cohorts of 3-6 patients receive escalating doses of resiquimod until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT).

* Step 3: Patients receive topical NY-ESO-1b peptide vaccine and topical resiquimod at the step 2 dose as in step 2.

Cohorts of 3-6 patients receive resiquimod to increasing amounts of surface area until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT.

Blood is drawn at baseline and periodically during study treatment and observation. Samples are analyzed by flow cytometry, monoclonal antibody staining, ELISPOT, and ELISA.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior diagnosis of melanoma meeting the following criteria:

  * Stage II-IV disease
  * Complete resection of disease
  * No current evidence of disease
* HLA-A2 positive
* No known standard therapy for disease that is potentially curative or proven capable of extending life expectancy exists

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 75,000/mm³
* AST ≤ 3 times upper limit of normal
* No uncontrolled or current infection
* No known allergy to vaccine or adjuvant components
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known immune deficiency

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy and recovered
* More than 4 weeks since prior biologic therapy
* No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number and severity of hematologic and non-hematologic toxicities | 4 weeks
Toxicity profile of each dose level | 4 weeks
Percent of patients who mount an immune response | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States